CLINICAL TRIAL: NCT02926911
Title: Comparing an Operation to Monitoring, With or Without Endocrine Therapy (COMET) Trial For Low Risk DCIS: A Phase III Prospective Randomized Trial
Brief Title: Comparing an Operation to Monitoring, With or Without Endocrine Therapy (COMET) Trial For Low Risk DCIS
Acronym: COMET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: Duke University (Other); Dana-Farber Cancer Institute (Other); New York University (Other); Washington University School of Medicine (Other); Patient-Centered Outcomes Research Institute (Other); M.D. Anderson Cancer Center (Other); Rising Tide Foundation (Other); Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFT-25
Record Dates: First submitted 2016-09-19; First posted 2016-10-06 (Estimated); Results first posted 2025-06-24 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-01

CONDITIONS: DCIS; Ductal Carcinoma in Situ
Keywords: Ductal Carcinoma
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Carcinoma, Ductal | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery (Active Comparator): DCIS - Surgery +/- radiation choice for endocrine therapy (MMG q 12 months x 5 years usual care for recurrent disease)
  Interventions: Other: Surgery
- Active Monitoring (Experimental): DCIS - Choice for endocrine therapy (MMG q 6 months x 5 years GCC for invasive progression)
  Interventions: Other: Active Monitoring

INTERVENTIONS:
Other: Surgery — Surgery +/- radiation choice for endocrine therapy
  Arms: Surgery
Other: Active Monitoring — Choice for endocrine therapy
  Arms: Active Monitoring

SUMMARY:
This study looks at the risks and benefits of active monitoring (AM) compared to surgery in the setting of a pragmatic prospective randomized trial for low risk DCIS. Our overarching hypothesis is that management of low-risk Ductal Carcinoma in Situ (DCIS) using an AM approach does not yield inferior cancer or quality of life outcomes compared to surgery.

DETAILED DESCRIPTION:
Overdiagnosis and overtreatment resulting from mammographic screening have been estimated to be as high as 1 in 4 patients diagnosed with breast cancer although the absence of standard definitions for measuring overdiagnosis has led to much uncertainty around this estimate. The national health care expenditure resulting from false positive mammograms and breast cancer overdiagnosis has been estimated to approach $4 billion annually. There is general consensus that much of this burden derives from the treatment of DCIS; for those estimated 40,000 women per year whose DCIS may never have progressed even without treatment, medical intervention can only harm. In those women who undergo surgical management of DCIS, there is risk of developing persistent pain at the surgical site, with estimates ranging from 25-68%. Importantly, persistent pain after lumpectomy may be as prevalent as that after total mastectomy. Persistent postsurgical pain is rated by patients as the most troubling symptom, leading to disability and psychological distress, and is often resistant to management. Although prospective population-based data have demonstrated significant patient and surgical focus on pain with remarkably high levels of chronic pain 4 and 9 months after breast surgery, much of these data have been collected in women with invasive cancer, with little data directly relevant to patients with DCIS.

The overarching hypothesis of the study is that management of low-risk DCIS using an active monitoring (AM) approach does not yield inferior cancer or quality of life outcomes compared to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unilateral, bilateral, unifocal, multifocal, or multicentric DCIS without invasive breast cancer (date of diagnosis defined as the date of the first pathology report that diagnosed the patient with DCIS) OR: atypia verging on DCIS OR: DCIS + LCIS (mix and/or separate locations in the same breast)
* A patient who has had a lumpectomy or partial mastectomy with margins positive for DCIS (i.e. <2mm/ink on tumor) as part of their treatment for a current DCIS diagnosis is also eligible (post-excision bilateral mammogram required at enrollment to establish a new baseline)
* No previous DCIS or invasive breast cancer in ipsilateral breast 5 years prior to current DCIS diagnosis
* 40 years of age or older at time of DCIS diagnosis
* ECOG performance status 0 or 1
* No contraindication for surgery
* Baseline imaging (must include dimensions):

  * Unilateral DCIS: contralateral normal mammogram ≤ 6 months of registration and ipsilateral breast imaging ≤ 120 days of registration (must include ipsilateral mammogram; can also include ultrasound or breast MRI)
  * Bilateral DCIS: bilateral breast imaging ≤ 120 days of registration (must include bilateral mammogram; can also include ultrasound or breast MRI)
  * DCIS s/p lumpectomy: post excision mammogram on side of excision ≤ 60 days of registration
* Pathologic criteria:

  * Any grade I DCIS (irrespective of necrosis/comedonecrosis)
  * Any grade II DCIS (irrespective of necrosis/comedonecrosis)
  * Absence of invasion or microinvasion
  * Diagnosis of DCIS confirmed on core needle biopsy, vacuum-assisted or surgery ≤ 120 days of registration
  * ER(+) and/or PR(+) by IHC (≥ 10% staining or Allred score ≥ 4) unless atypia verging on DCIS in which case biomarker criterion does not apply
  * HER2 0, 1+, or 2+ by IHC if HER2 testing is performed
* Histology slides reviewed and agreement between two clinical pathologists (not required to be at same institution) that pathology fulfills COMET eligibility criteria. In cases of disagreement between the two pathology reviews about whether or not a case fulfills the eligibility criteria, a third pathology review will be required.
* At least two sites of biopsy for those cases where individual mammographic extent of calcifications exceeds 4 cm, with second biopsy benign or both sites fulfilling pathology eligibility criteria (ER/PR testing required for second biopsy)
* Amenable to follow up examinations
* Ability to read, understand and evaluate study materials and willingness to sign a written informed consent document
* Reads and speaks Spanish or English

Exclusion Criteria:

* Male DCIS
* Grade III DCIS
* Concurrent diagnosis of invasive or microinvasive breast cancer in either breast
* Documented mass on examination or mass/hypoechoic area on imaging at site of DCIS prior to biopsy yielding diagnosis of DCIS, with exception of: subsequent lumpectomy or partial mastectomy (with positive DCIS margins i.e. <2mm/ink on tumor) followed by a post-surgery MMG; fibroadenoma at a distinct/separate site from site of DCIS; or diagnosis of mass/hypoechoic area as a cyst or a papilloma. In cases of uncertainty about whether the mass was present on physical examination prior to biopsy, the following criteria should be applied: if mammogram noting abnormal findings is diagnostic MMG = symptomatic/if mammogram noting abnormal findings is screening MMG = asymptomatic. If a patient has a mass on imaging that is biopsied (worked-up) and does not show invasive breast cancer, they are eligible. If a patient has a mass on initial MMG that is not seen on subsequent MMG, they are eligible (if initial mass occurred due to additional work-up).
* Any color/bloody nipple discharge (ipsilateral breast)
* Mammographic finding of BIRADS 4 or greater within 6 months prior to registration at site of breast other than that of known DCIS, without pathologic assessment
* Use of investigational cancer agents within 6 weeks prior to diagnosis of DCIS
* Any serious and/or unstable pre-existing medical, psychiatric, or other existing condition that would prevent compliance with the trial or consent process
* Pregnancy. If a woman has been confirmed as pregnant, she will not be eligible to take part in the trial. If she suspects there is a chance that she may be pregnant, a pregnancy test should be undertaken, although a pregnancy test for all women of child-bearing potential is not mandatory. In addition, if a woman becomes pregnant once registered to the trial, she can continue to be followed (endocrine therapy is not a mandatory requirement of the study)
* Documented history of prior tamoxifen, aromatase inhibitor, or raloxifene use in the 6 months prior to registration
* Current use of exogenous hormones (i.e. oral progesterone)

Ages: 40 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 997 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2030-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shelley Hwang, MD, MPH, Principal Investigator — Duke University; Ann Partridge, MD, MPH, Study Chair — Dana-Farber Cancer Institute; Alastair Thompson, MD, Study Chair — Baylor College of Medicine
Locations (139):
- United States (139):
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic, Phoenix, Arizona
  - City of Hope, Duarte, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sharp Memorial Hospital, San Diego, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - Colorado Cancer Research Program, Denver, Colorado
  - Saint Joseph Hospital- Cancer Centers of Colorado, Lafayette, Colorado
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Memorial Healthcare System, Hollywood, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kootenai Health, Post Falls, Idaho
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Medical Oncology and Hematology Associates - Des Moines, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - St. Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center Cancer Care, Brewer, Maine
  - Maine Center for Cancer Medicine-Scarborough, Scarborough, Maine
  - New England Cancer Specialists, Scarborough, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland - Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Cancer Research Consortium of West Michigan, Grand Rapids, Michigan
  - Beaumont NCORP, Royal Oak, Michigan
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro MN Community Oncology Research Consortium (MMCORC), Saint Louis Park, Minnesota
  - Washington University - Siteman Cancer Center, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic, Billings, Montana
  - Bozeman Health, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New Hampshire Oncology Hematology PA, Hooksett, New Hampshire
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Atlantic Health System / Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York-Presbyterian Weill Cornell Medical Center, New York, New York
  - Mount Sinai Hospital, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore-Einstein Center for Cancer Care at Montefiore Medical Park, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Novant Health Breast Surgery - Greensboro, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Carolina East Medical Center, New Bern, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Strecker Cancer Center - Belpre, Belpre, Ohio
  - Dayton Physicians-Miami Valley Hospital South, Centerville, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology & Hematology INC, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - MidOhio Oncology Hematology, Mark H. Zangmeister Center, Columbus, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Dayton Physicians-Miami Valley Hospital North, Dayton, Ohio
  - Grady Hospital, Delaware, Ohio
  - OhioHealth Grady - Delaware Health Center, Delaware, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Dayton Physicians-Atrium, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - St. Ann's Hospital, Westerville, Ohio
  - St. Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Health Care System, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma, Lawton, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - WellSpan Health York Cancer Center, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Georgetown Hospital System, Georgetown, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Baptist Cancer Care, Memphis, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Doctors Hospital of Laredo, Laredo, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - The University of Vermont Medical Center, Burlington, Vermont
  - West Virginia University Medicine, Morgantown, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Overlake Hospital Medical Center, Bellevue, Washington
  - ThedaCare Regional Cancer Center -Appleton, Appleton, Wisconsin
  - Aurora Health Care, Aurora Cancer Care, Burlington, Wisconsin
  - Aurora Health Center - Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care, Germantown Health Center, Germantown, Wisconsin
  - Aurora Health Care, Aurora Cancer Care, Grafton, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - BayCare Aurora LLC, Aurora Cancer Care, Green Bay, Wisconsin
  - Aurora Health Care, Aurora Cancer Care, Kenosha, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Aurora Bay Area Medical Group - Cancer Care Clinic, Marinette, Wisconsin
  - Aurora Health Care, Aurora Cancer Care, Marinette, Wisconsin
  - Aurora Health Care, Aurora Cancer Care, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic of Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Health Care, Aurora Cancer Care, Oshkosh, Wisconsin
  - Aurora Health Care, Aurora Cancer Care, Racine, Wisconsin
  - Aurora Health Care, Aurora Cancer Care, Sheboygan, Wisconsin
  - Aurora Health Care, Aurora Cancer Care, Summit, Wisconsin
  - Aurora Health Care, Aurora Cancer Care, Two Rivers, Wisconsin
  - Aurora Health Care, Aurora Cancer Care, Wauwatosa, Wisconsin
  - Aurora Health Care, Aurora Cancer Care, West Allis, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient medical information both, associated with biologic specimens or not, is confidential and may only be disclosed to third parties as permitted by the Informed Consent Form (ICF) (or separate authorization for use and disclosure of personal health information) which has been signed by the patient, unless permitted or required by law. Data derived from biologic specimen analysis on individual patients will in generally not be provided to study investigators unless a request for research use is granted. The overall results of any research conducted using biologic specimens will be available in accordance with the effective Alliance Foundation Trial (AFT) policy on study data publication.
Time Frame: Data will become available July 2023, no end date.
Access Criteria: following a formal request by an investigator to and approval from AFT

REFERENCES:
- [Background] Ernster VL, Ballard-Barbash R, Barlow WE, Zheng Y, Weaver DL, Cutter G, Yankaskas BC, Rosenberg R, Carney PA, Kerlikowske K, Taplin SH, Urban N, Geller BM. Detection of ductal carcinoma in situ in women undergoing screening mammography. J Natl Cancer Inst. 2002 Oct 16;94(20):1546-54. doi: 10.1093/jnci/94.20.1546. PMID 12381707
- [Background] Erbas B, Provenzano E, Armes J, Gertig D. The natural history of ductal carcinoma in situ of the breast: a review. Breast Cancer Res Treat. 2006 May;97(2):135-44. doi: 10.1007/s10549-005-9101-z. Epub 2005 Dec 1. PMID 16319971
- [Background] Ozanne EM, Shieh Y, Barnes J, Bouzan C, Hwang ES, Esserman LJ. Characterizing the impact of 25 years of DCIS treatment. Breast Cancer Res Treat. 2011 Aug;129(1):165-73. doi: 10.1007/s10549-011-1430-5. Epub 2011 Mar 9. PMID 21390494
- [Background] Nystrom L, Rutqvist LE, Wall S, Lindgren A, Lindqvist M, Ryden S, Andersson I, Bjurstam N, Fagerberg G, Frisell J, et al. Breast cancer screening with mammography: overview of Swedish randomised trials. Lancet. 1993 Apr 17;341(8851):973-8. doi: 10.1016/0140-6736(93)91067-v. PMID 8096941
- [Derived] Partridge AH, Hyslop T, Rosenberg SM, Bennett AV, Drier S, Jonsson M, Shimada A, Li Y, Li Y, Lynch T, Frank E, Collyar D, Basila D, Pinto D, Weiss A, Wolf A, Norris K, Witten M, Boisvert M, Giuliano A, Larson KE, Yost K, McAuliffe PF, Krie A, Tamirisa N, Darai S, Carey L, Thompson A, Hwang ES; COMET Study Consortium. Patient-Reported Outcomes for Low-Risk Ductal Carcinoma In Situ: A Secondary Analysis of the COMET Randomized Clinical Trial. JAMA Oncol. 2025 Mar 1;11(3):300-309. doi: 10.1001/jamaoncol.2024.6556. PMID 39665588
- [Derived] Hwang ES, Hyslop T, Lynch T, Ryser MD, Weiss A, Wolf A, Norris K, Witten M, Grimm L, Schnitt S, Badve S, Factor R, Frank E, Collyar D, Basila D, Pinto D, Watson MA, West R, Davies L, Donovan JL, Shimada A, Li Y, Li Y, Bennett AV, Rosenberg S, Marks J, Winer E, Boisvert M, Giuliano A, Larson KE, Yost K, McAuliffe PF, Krie A, Tamirisa N, Carey LA, Thompson AM, Partridge AH; COMET Study Investigators. Active Monitoring With or Without Endocrine Therapy for Low-Risk Ductal Carcinoma In Situ: The COMET Randomized Clinical Trial. JAMA. 2025 Mar 18;333(11):972-980. doi: 10.1001/jama.2024.26698. PMID 39665585
- [Derived] Ozanne EM, Maves K, Tramontano AC, Lynch T, Thompson A, Partridge A, Frank E, Collyar D, Basila D, Pinto D, Hyslop T, Ryser MD, Rosenberg S, Hwang ES, Punglia RS. Impact of an online decision support tool for ductal carcinoma in situ (DCIS) using a pre-post design (AFT-25). Breast Cancer Res. 2024 Sep 17;26(1):134. doi: 10.1186/s13058-024-01891-w. PMID 39289750
- [Derived] Hwang ES, Hyslop T, Lynch T, Frank E, Pinto D, Basila D, Collyar D, Bennett A, Kaplan C, Rosenberg S, Thompson A, Weiss A, Partridge A. The COMET (Comparison of Operative versus Monitoring and Endocrine Therapy) trial: a phase III randomised controlled clinical trial for low-risk ductal carcinoma in situ (DCIS). BMJ Open. 2019 Mar 12;9(3):e026797. doi: 10.1136/bmjopen-2018-026797. PMID 30862637

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Monitoring: DCIS - Choice for endocrine therapy (MMG q 6 months x 5 years GCC for invasive progression) >
  > Active Monitoring: Choice for endocrine therapy
- Surgery: DCIS - Surgery +/- radiation choice for endocrine therapy (MMG q 12 months x 5 years usual care for recurrent disease) >
  > Surgery: Surgery +/- radiation choice for endocrine therapy
Period: Overall Study
Arm/Group | Active Monitoring | Surgery
Started | 497 | 498
Completed | 484 | 473
Not Completed | 13 | 25

BASELINE CHARACTERISTICS:
Groups:
- Active Monitoring: DCIS - Choice for endocrine therapy (MMG q 6 months x 5 years GCC for invasive progression)>
  > Active Monitoring: Choice for endocrine therapy
- Surgery: DCIS - Surgery +/- radiation choice for endocrine therapy (MMG q 12 months x 5 years usual care for recurrent disease)>
  > Surgery: Surgery +/- radiation choice for endocrine therapy
- Total: Total of all reporting groups
Arm/Group | Active Monitoring | Surgery | Total
Number analyzed (Participants) | 484 | 473 | 957
Age, Customized [Count of Participants; unit: Participants]
  <55 | 112 | 114 | 226
  55-65 | 164 | 164 | 328
  >65 | 208 | 195 | 403
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 484 | 473 | 957
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 17 | 51
  Not Hispanic or Latino | 438 | 440 | 878
  Unknown or Not Reported | 12 | 16 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 23 | 23 | 46
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 80 | 70 | 150
  White | 359 | 359 | 718
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 18 | 15 | 33
DCIS laterality at diagnosis [Count of Participants; unit: Participants]
  Left | 247 | 235 | 482
  Right | 233 | 236 | 469
  Bilateral | 4 | 2 | 6
DCIS grade at diagnosis [Count of Participants; unit: Participants] — A DCIS diagnosis is categorized as low-grade (grade I), intermediate grade (grade II), or high-grade (grade III). The higher the grade, the more abnormal the nuclei and the more aggressive and fast-growing the cancer cells.
  Participants
    1 | 125 | 127 | 252
    2 | 359 | 346 | 705
DCIS estrogen receptor positive at diagnosis [Count of Participants; unit: Participants] | 473 | 467 | 940
DCIS progesterone receptor status at diagnosis [Count of Participants; unit: Participants] — Population: Some patients' receptor status was not collected
  Participants
    Positive: number analyzed (Participants) | 405 | 411 | 816
    Positive | 364 | 359 | 723
    Negative: number analyzed (Participants) | 405 | 411 | 816
    Negative | 41 | 52 | 93
DCIS ERBB2 status at diagnosis [Count of Participants; unit: Participants] — 0 and 1+ are both HER2-negative. Lower score is better. Population: Some patients' status was not collected
  Participants
    0: number analyzed (Participants) | 4 | 8 | 12
    0 | 1 | 3 | 4
    1+: number analyzed (Participants) | 4 | 8 | 12
    1+ | 3 | 5 | 8
Premenopausal/perimenopausal [Count of Participants; unit: Participants] | 90 | 92 | 182
ECOG performance status score [Count of Participants; unit: Participants] — 0: Fully active, able to carry out normal activities without restriction.
  1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  Participants
    0 | 431 | 410 | 841
    1 | 53 | 63 | 116
Comorbidities [Count of Participants; unit: Participants] | 284 | 256 | 540
Total No. of comorbidities [Count of Participants; unit: Participants] — Population: Analysis population is subset of patients who had any comorbidity
  Participants
    0: number analyzed (Participants) | 432 | 431 | 863
    0 | 148 | 175 | 323
    1: number analyzed (Participants) | 432 | 431 | 863
    1 | 137 | 124 | 261
    2: number analyzed (Participants) | 432 | 431 | 863
    2 | 58 | 55 | 113
    3: number analyzed (Participants) | 432 | 431 | 863
    3 | 34 | 27 | 61
    4: number analyzed (Participants) | 432 | 431 | 863
    4 | 14 | 11 | 25
    5+: number analyzed (Participants) | 432 | 431 | 863
    5+ | 41 | 39 | 80

OUTCOME MEASURES:

1. Primary Outcome: Proportion of New Diagnoses of Ipsilateral Invasive Cancer in Surgery and AM Arms at 2 Years of Follow up
Description: To compare the number of patients that develop ipsilateral invasive cancer that received surgery to the number of patients that were placed on active monitoring after 2 years of follow-up
Time Frame: At 2 years follow-up
Measure: Number (95% Confidence Interval); unit: "percentage of participants
Arm/Group | Active Monitoring | Surgery
Number analyzed (Participants) | 484 | 473
"percentage of participants | 4.2 [2.31 to 6.00] | 5.9 [3.71 to 8.04]

2. Secondary Outcome: Quality of Life (QOL)
Description: Measured by Short Form (SF)-36
Time Frame: Baseline, 6 months, 1 year, and once a year (years 2 through 5)
Reporting Status: Not Posted

3. Secondary Outcome: Psychological Outcomes
Description: Measured by five dimensions questionnaire (EQ-5D)
Time Frame: Baseline, 6 months, 1 year, and once a year (years 2 through 5)
Reporting Status: Not Posted

4. Secondary Outcome: Generalized Anxiety
Description: Measured by the State Trait Anxiety Inventory (STAI) scale
Time Frame: Baseline, 6 months, 1 year, and once a year (years 2 through 5)
Reporting Status: Not Posted

5. Secondary Outcome: Generalized Depression
Description: Measured by the Center for Epidemiologic Studies Depression Scale (CES-D) 10
Time Frame: Baseline, 6 months, 1 year, and once a year (years 2 through 5)
Reporting Status: Not Posted

6. Secondary Outcome: Coping
Description: Coping evaluated using the Brief COPE, a shortened form of the COPE Inventory, inclusive of 28 items (14 subscales).
Time Frame: Baseline
Reporting Status: Not Posted

7. Secondary Outcome: Intolerance of Uncertainty
Description: Assessment of feelings of uncertainty using the Intolerance of Uncertainty Scale (Short-form), which has been used in studies of active monitoring in the prostate cancer setting.
Time Frame: Baseline and at 2 years
Reporting Status: Not Posted

8. Secondary Outcome: Mastectomy Rate
Description: To compare the impact of surgery vs. AM on the number of mastectomies performed in patients with DCIS
Time Frame: 2, 5, and 7 year follow-up
Reporting Status: Not Posted

9. Secondary Outcome: Breast Conservation Rate
Description: To compare the impact of surgery vs. AM on the number of breast conservation surgeries performed in patients with DCIS
Time Frame: 2, 5, and 7 year follow-up
Reporting Status: Not Posted

10. Secondary Outcome: Contralateral Invasive Cancer Rate
Description: To compare the impact of surgery vs. AM on the rate of development of contralateral invasive cancer in patients with DCIS
Time Frame: 2, 5, and 7 year follow-up
Reporting Status: Not Posted

11. Secondary Outcome: Overall Survival Rate
Description: To compare the impact of surgery vs. AM on the overall survival rate in patients with DCIS
Time Frame: 2, 5, and 7 year follow-up
Reporting Status: Not Posted

12. Secondary Outcome: Breast Cancer Specific Survival Rate
Description: To compare the impact of surgery vs. AM on the breast cancer specific survival rate in patients with DCIS
Time Frame: 2, 5, and 7 year follow-up
Reporting Status: Not Posted

13. Secondary Outcome: Ipsilateral Invasive Cancer Rate in Surgery Arm at 5 and 7 Year Follow-up
Description: To determine the number of DCIS patients in the surgery arm that develop ipsilateral invasive cancer
Time Frame: 5 and 7 year follow-up
Reporting Status: Not Posted

14. Secondary Outcome: Ipsilateral Invasive Cancer Rate in AM Arm
Description: To determine the number of DCIS patients in the AM arm that develop ipsilateral invasive cancer
Time Frame: 5 and 7 year follow-up
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Breast MRI Utilization Rate
Description: Determine the rate of use of breast MRI imaging compared to use of other breast imaging techniques
Time Frame: 2, 5, and 7 year follow-up
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Breast Biopsy Rate
Description: Determine the rate of biopsies performed during follow-up of patients with DCIS
Time Frame: 2, 5, and 7 year follow-up
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Radiation Rate
Description: Determine the rate of the performance of radiation therapy on patients with DCIS
Time Frame: 2, 5, and 7 year follow-up
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Chemotherapy Rate
Description: Determine the rate of the use of chemotherapy on patients with DCIS
Time Frame: 2, 5, and 7 year follow-up
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Self-reported Co-morbidity
Description: Self-reported diary
Time Frame: 6 months, 1 year, and once a year (years 2 through 5)
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Adherence to Hormonal Therapy
Description: Evaluated with a drug diary
Time Frame: 6 months, 1 year, and once a year (years 2 through 5)
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Symptoms
Description: A modified 19-item version of the Breast Cancer Prevention Trial (BCPT) Symptom Checklist will evaluate commonly reported menopausal symptoms
Time Frame: Baseline, 6 months, 1 year, and once a year (years 2 through 5)
Reporting Status: Not Posted

22. Other Pre Specified Outcome: General Pain
Description: Evaluated with the Brief Pain Inventory, a well-validated general measure of pain and disability worst pain, least pain, and interference
Time Frame: Baseline, 6 months, 1 year, and once a year (years 2 through 5)
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Breast Specific Pain
Description: Breast specific pain will be measured by the Breast Cancer Pain Questionnaire (BCPQ); the BCPQ includes assessment of pain severity, pain frequency (how many days/week), and pain location (breast, arm, side, axilla), from which a Pain Burden Index (PBI) can be calculated
Time Frame: Baseline, 6 months, 1 year, and once a year (years 2 through 5)
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Body Image
Description: Body image will be evaluated by the Breast-Questionnaire, a validated instrument to evaluate outcomes following surgery, will be used to evaluate satisfaction with body image
Time Frame: Baseline, 6 months, 1 year, and once a year (years 2 through 5)
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Decisional Regret
Description: The Decision Regret Scale will measure how women perceived their DCIS treatment decision. The SURE scale, which is composed of four items from the Decisional Conflict Scale will be used to measure patients' uncertainty about which treatment to choose and factors contributing to uncertainty (feeling uninformed, unclear values, and unsupported in decision-making).
Time Frame: Years 1 through 5
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Knowledge
Description: DCIS and breast cancer knowledge will be measured with items adapted from the Breast Cancer Surgery Decision Quality Instrument (BCS-DQI) as well as questions developed specifically for a study that assessed DCIS knowledge and risk perceptions. The investigators will assess risk perceptions in women with DCIS using questions developed by Lerman and Croyle that will measure risk perceptions in relation to psychosocial outcomes in women with DCIS
Time Frame: Baseline and 2 years
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Risk Perceptions
Description: Measured by the Breast Cancer Surgery Decision Quality Instrument (BCS-DQI)
Time Frame: Baseline and 2 years
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Communication With Physicians
Description: To assess communication with physicians about DCIS management options, the investigators will adapt items used in a prior study of surgical decision-making, including the extent to which their physician talked to them about AM vs. surgery. Additionally the investigators will ask about sources of information for the management of their DCIS
Time Frame: Baseline
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Financial Burden
Description: The investigators will adapt items from the National Health Interview Survey and the Cancer Outcomes Research and Surveillance (CanCORS) Study to assess financial burden. The investigators will also ask women to Cancer Care estimate out of pocket expenses attributed to their DCIS diagnosis.
Time Frame: 6 months
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Employment Status
Description: Employment status will be assessed using a measure that is being added to the Alliance Patient Questionnaire as it has been tested and validated in breast cancer populations.
Time Frame: Baseline, 6 months, year 1, and once a year (years 1 through 5)
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Concerns About Future Breast Events
Description: Four items from the Quality of Life in Adult Cancer Survivors (QLACS) scale will be adapted to evaluate frequency (1=never; 7=always) of worries about DCIS, including concerns about future breast events and death from DCIS
Time Frame: Baseline and 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Active Monitoring | Surgery
All-Cause Mortality (participants affected / at risk) | 11/484 | 8/473
Serious Adverse Events (participants affected / at risk) | 11/484 | 8/473
Other Adverse Events (participants affected / at risk) | 378/484 | 351/473
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Monitoring (N=484) | Surgery (N=473)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 6 (6) | 4 (4)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Monitoring (N=484) | Surgery (N=473)
Anemia (Blood and lymphatic system disorders) | 8 (12) | 7 (10)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Spleen disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 3 (8)
Aortic valve disease (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 1 (2) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (2) | 1 (2)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 2 (2)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (3) | 0 (0)
Mobitz (type) II atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Mobitz type I (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 5 (6) | 3 (3)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 4 (4) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 2 (3) | 4 (5)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 2 (4) | 3 (6)
Tinnitus (Ear and labyrinth disorders) | 1 (5) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (2) | 1 (1)
Hypothyroidism (Endocrine disorders) | 5 (7) | 2 (2)
Blurred vision (Eye disorders) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 3 (3) | 2 (2)
Dry eye (Eye disorders) | 4 (7) | 1 (2)
Eye disorders - Other, specify (Eye disorders) | 1 (4) | 2 (4)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Floaters (Eye disorders) | 1 (4) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Retinal vascular disorder (Eye disorders) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 1 (2) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (8) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 6 (9) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 0 (0)
Esophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 (13) | 3 (4)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1) | 1 (4)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 50 (117) | 43 (77)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 4 (4)
Chills (General disorders) | 2 (2) | 2 (9)
Edema limbs (General disorders) | 10 (14) | 8 (11)
Fatigue (General disorders) | 27 (62) | 29 (46)
Fever (General disorders) | 22 (30) | 17 (22)
Flu like symptoms (General disorders) | 4 (8) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 8 (10) | 3 (3)
Localized edema (General disorders) | 2 (3) | 3 (5)
Non-cardiac chest pain (General disorders) | 1 (1) | 3 (3)
Pain (General disorders) | 7 (13) | 10 (12)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 2 (2)
Allergic reaction (Immune system disorders) | 16 (37) | 12 (17)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Breast infection (Infections and infestations) | 1 (1) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 2 (3)
Conjunctivitis (Infections and infestations) | 1 (2) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 9 (11) | 9 (9)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (2) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 3 (6) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 5 (5) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 7 (11)
Vaginal infection (Infections and infestations) | 4 (5) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 9 (10)
Fracture (Injury, poisoning and procedural complications) | 29 (50) | 21 (24)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 4 (7) | 2 (3)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (4) | 1 (1)
Alkaline phosphatase increased (Investigations) | 3 (5) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 80 (216) | 76 (175)
Creatinine increased (Investigations) | 2 (4) | 2 (2)
Investigations - Other, specify (Investigations) | 1 (1) | 3 (12)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 3 (3)
Weight gain (Investigations) | 6 (8) | 10 (17)
Weight loss (Investigations) | 5 (12) | 3 (7)
White blood cell decreased (Investigations) | 3 (3) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 4 (7) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (13) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 2 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Obesity (Metabolism and nutrition disorders) | 9 (20) | 8 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 178 (596) | 167 (528)
Arthritis (Musculoskeletal and connective tissue disorders) | 12 (20) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 11 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 4 (6) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 8 (10) | 16 (39)
Myalgia (Musculoskeletal and connective tissue disorders) | 88 (234) | 88 (235)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 92 (296) | 98 (280)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (12) | 5 (5)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (16) | 10 (10)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 3 (4) | 2 (3)
Concentration impairment (Nervous system disorders) | 3 (4) | 0 (0)
Dizziness (Nervous system disorders) | 9 (11) | 9 (15)
Dysarthria (Nervous system disorders) | 2 (2) | 0 (0)
Dysesthesia (Nervous system disorders) | 2 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Glossopharyngeal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 12 (24) | 10 (15)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 2 (2) | 5 (10)
Memory impairment (Nervous system disorders) | 4 (11) | 6 (9)
Muscle weakness right-sided (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Oth spec (Nervous system disorders) | 2 (3) | 5 (7)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (4)
Paresthesia (Nervous system disorders) | 2 (3) | 4 (5)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 2 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (13) | 9 (17)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (2)
Vasovagal reaction (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 9 (12) | 7 (7)
Confusion (Psychiatric disorders) | 1 (1) | 1 (2)
Depression (Psychiatric disorders) | 10 (18) | 5 (7)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 14 (16) | 6 (22)
Libido decreased (Psychiatric disorders) | 2 (2) | 1 (1)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 2 (3) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (1) | 3 (4)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 4 (5) | 6 (12)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 15 (24) | 12 (24)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 2 (3) | 4 (12)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Menorrhagia (Reproductive system and breast disorders) | 3 (6) | 2 (3)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 6 (7) | 4 (6)
Vaginal discharge (Reproductive system and breast disorders) | 7 (23) | 6 (14)
Vaginal dryness (Reproductive system and breast disorders) | 8 (16) | 9 (28)
Vaginal hemorrhage (Reproductive system and breast disorders) | 5 (5) | 2 (2)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (11) | 8 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (16) | 9 (21)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (17)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (5) | 4 (4)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 6 (9) | 7 (13)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Menopause (Social circumstances) | 1 (5) | 0 (0)
Social circumstances - Other, specify (Social circumstances) | 0 (0) | 3 (5)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 8 (16) | 2 (3)
Hematoma (Vascular disorders) | 1 (4) | 0 (0)
Hot flashes (Vascular disorders) | 208 (688) | 193 (723)
Hypertension (Vascular disorders) | 229 (855) | 198 (731)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 3 (5)
Superficial thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 4 (6) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT02926911/Prot_SAP_000.pdf